CLINICAL TRIAL: NCT00772824
Title: Study of the Effect of Glutamine Supplementation on Chemotherapy Induced Toxicities in Breast Cancer Patients- A Prospective, Randomised, Single Blind, Three Arm, Phase Four Prevention Trial
Brief Title: Study of the Effect of Glutamine Supplementation on Chemotherapy Induced Toxicities in Breast Cancer Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Banaras Hindu University (Other)
Responsible Party: Principal Investigator, Manoj Pandey, Professor, Surgical Oncology, Banaras Hindu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GLU_07
Record Dates: First submitted 2008-10-14; First posted 2008-10-15 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Chemotherapy; Epirubicin; Glutamine; FEC chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Glutamine

STUDY DESIGN:
Intervention Model Description: Case Control
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (No Intervention): 10 patients (30 cycles) of chemotherapy will receive placebo
- 2 (Active Comparator): Intravenous glutamine
  Interventions: Dietary Supplement: IV Glutamine
- 3 (Experimental): Oral Glutamine
  Interventions: Dietary Supplement: Glutamine

INTERVENTIONS:
Dietary Supplement: Glutamine — 2g/kg body weight twice daily in divided doses for 5 days
  Arms: 3
Dietary Supplement: IV Glutamine — 50 ml of 20% glutamine IV before chemotherapy
  Arms: 2

SUMMARY:
Glutamine, a non essential branched chain amino acid, is most important non toxic nitrogen carrier in body. It participates in variety of physiological functions. It is a major fuel source of enterocytes and is a substrate for gluconeogenesis in kidney, lymphocytes, and monocytes. It is also a nutrient in muscle protein metabolism in response to infection, inflammation and muscle trauma. The significance of glutamine to metabolic homeostasis becomes evident during periods of stress, when it becomes a conditionally essential amino acid. Role of glutamine as protective agent in hepato-biliary dysfunction, in maintaining mucosal integrity of the Gastrointestinal tract following its administration in patient with major bowel surgery as a supplement and part of TPN in critically ill patients and in patients of septicemia, is well established. However the role of glutamine supplementation in reducing or preventing chemotherapeutic agents induced toxicity in cancer patients is controversial.

ELIGIBILITY:
Inclusion Criteria:

* The patients > 18 years of age
* Histologically or cytologically proven breast cancer
* Receiving CEF chemotherapy cycles presently or in the past
* The patients who will give informed consent to participate in the study
* Patients must have sufficient organ and marrow function
* Stage 1 neuropathy, subclinical neuropathy, surgery induced neuropathy

Exclusion Criteria:

* Pregnancy
* Clinical/biochemical severe liver failure
* Clinical/biochemical severe renal dysfunction
* Refusal to participate in the study
* Patients who have received prior chemotherapy with paclitaxel.
* Patients who have neuropathy due to any known systemic or metabolic causes like diabetes, leprosy, nutritional deficiency induced (vit. B12) etc

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Reduction in toxicity | 3 weeks

SECONDARY OUTCOMES:
Serum level of creatinine kinase and LDH | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: R K Goel, MD, Principal Investigator — Institute of Medical Sciences
Locations (1):
- Sir Sunder Lal Hospital, Varanasi, Uttar Pradesh, India

REFERENCES:
- [Background] Bergstrom J, Furst P, Noree LO, Vinnars E. Intracellular free amino acid concentration in human muscle tissue. J Appl Physiol. 1974 Jun;36(6):693-7. doi: 10.1152/jappl.1974.36.6.693. No abstract available. PMID 4829908
- [Background] Lacey JM, Wilmore DW. Is glutamine a conditionally essential amino acid? Nutr Rev. 1990 Aug;48(8):297-309. doi: 10.1111/j.1753-4887.1990.tb02967.x. PMID 2080048
- [Background] Daniele B, Perrone F, Gallo C, Pignata S, De Martino S, De Vivo R, Barletta E, Tambaro R, Abbiati R, D'Agostino L. Oral glutamine in the prevention of fluorouracil induced intestinal toxicity: a double blind, placebo controlled, randomised trial. Gut. 2001 Jan;48(1):28-33. doi: 10.1136/gut.48.1.28. PMID 11115819
- [Background] Rubio IT, Cao Y, Hutchins LF, Westbrook KC, Klimberg VS. Effect of glutamine on methotrexate efficacy and toxicity. Ann Surg. 1998 May;227(5):772-8; discussion 778-80. doi: 10.1097/00000658-199805000-00018. PMID 9605669
- [Background] Satoh J, Tsujikawa T, Fujiyama Y, Bamba T. Nutritional benefits of enteral alanyl-glutamine supplementation on rat small intestinal damage induced by cyclophosphamide. J Gastroenterol Hepatol. 2003 Jun;18(6):719-25. doi: 10.1046/j.1440-1746.2003.03042.x. PMID 12753156
- [Background] van der Hulst RR, van Kreel BK, von Meyenfeldt MF, Brummer RJ, Arends JW, Deutz NE, Soeters PB. Glutamine and the preservation of gut integrity. Lancet. 1993 May 29;341(8857):1363-5. doi: 10.1016/0140-6736(93)90939-e. PMID 8098788
- [Background] Govindarajan R, Heaton KM, Broadwater R, Zeitlin A, Lang NP, Hauer-Jensen M. Effect of thalidomide on gastrointestinal toxic effects of irinotecan. Lancet. 2000 Aug 12;356(9229):566-7. doi: 10.1016/s0140-6736(00)02586-1. PMID 10950238
- [Background] Berthrong M. Pathologic changes secondary to radiation. World J Surg. 1986 Apr;10(2):155-70. doi: 10.1007/BF01658133. No abstract available. PMID 3705602
- [Background] Huang EY, Leung SW, Wang CJ, Chen HC, Sun LM, Fang FM, Yeh SA, Hsu HC, Hsiung CY. Oral glutamine to alleviate radiation-induced oral mucositis: a pilot randomized trial. Int J Radiat Oncol Biol Phys. 2000 Feb 1;46(3):535-9. doi: 10.1016/s0360-3016(99)00402-2. PMID 10701731
- [Background] Cao Y, Kennedy R, Klimberg VS. Glutamine protects against doxorubicin-induced cardiotoxicity. J Surg Res. 1999 Jul;85(1):178-82. doi: 10.1006/jsre.1999.5677. PMID 10383856
- [Background] Boyle FM, Wheeler HR, Shenfield GM. Amelioration of experimental cisplatin and paclitaxel neuropathy with glutamate. J Neurooncol. 1999 Jan;41(2):107-16. doi: 10.1023/a:1006124917643. PMID 10222430
- [Background] Vahdat L, Papadopoulos K, Lange D, Leuin S, Kaufman E, Donovan D, Frederick D, Bagiella E, Tiersten A, Nichols G, Garrett T, Savage D, Antman K, Hesdorffer CS, Balmaceda C. Reduction of paclitaxel-induced peripheral neuropathy with glutamine. Clin Cancer Res. 2001 May;7(5):1192-7. PMID 11350883